CLINICAL TRIAL: NCT02392091
Title: Renal Tubular Acidosis is Highly Prevalent in Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Richard Brunner, MD, Dr, Medical University of Vienna
Other Study IDs: RTA01
Record Dates: First submitted 2015-03-12; First posted 2015-03-18 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Acidosis, Renal Tubular
MeSH Terms: conditions — Acidosis, Renal Tubular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- critically ill patients: critically ill patients at the age ≥18, expected to stay in the ICU for ≥24h, with the clinical necessity for a urinary catheter and the absence of anuria

SUMMARY:
The aim of this study was to investigate the prevalence, type, and possible risk factors of RTA in critically ill patients using a physical-chemical approach.

DETAILED DESCRIPTION:
Hyperchloremic acidosis is frequent in critically ill patients. Renal tubular acidosis (RTA) may contribute to acidemia in the state of hyperchloremic acidosis, but the prevalence of RTA has never been studied in critically ill patients. Therefore, we aimed to investigate the prevalence, type, and possible risk factors of RTA in critically ill patients using a physical-chemical approach.

This prospective, observational trial was conducted in a medical ICU of a university hospital. 100 consecutive critically ill patients at the age ≥18, expected to stay in the ICU for ≥24h, with the clinical necessity for a urinary catheter and the absence of anuria were included.

Base excess subset calculation based on a physical-chemical approach on the first seven days after ICU admission was used to compare the effects of free water, chloride, albumin, and unmeasured anions on the standard base excess. Calculation of the urine osmolal gap (UOG) - as an approximate measure of the unmeasured urine cation ammonium - served as determinate between renal and extra-renal bicarbonate loss in the state of hyperchloremic acidosis.

ELIGIBILITY:
Inclusion Criteria:

* admitted to the medical ICU of the Div. of Gastroenterology & Hepatology of the Medical University of vienna
* age ≥18
* expectancy to stay in the ICU ≥24hours
* clinical necessity for a urinary catheter

Exclusion Criteria:

* anuria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients from a medical ICU
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2011-04; Primary Completion 2011-10 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
renal-tubular acidosis | up to 7 days after ICU admission
  Diagnosis of renal-tubular acidosis in critically ill patients within 7 days after ICU admission.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Brunner, MD, Principal Investigator — Medical University of Vienna

REFERENCES:
- [Derived] Brunner R, Drolz A, Scherzer TM, Staufer K, Fuhrmann V, Zauner C, Holzinger U, Schneeweiss B. Renal tubular acidosis is highly prevalent in critically ill patients. Crit Care. 2015 Apr 6;19(1):148. doi: 10.1186/s13054-015-0890-0. PMID 25888397